CLINICAL TRIAL: NCT00193245
Title: A Randomized Trial of Oral Topotecan Versus Docetaxel in Second-Line Treatment of Non-Small Cell Lung Cancer
Brief Title: Oral Topotecan Versus Docetaxel in Second-Line Treatment of Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: AstraZeneca (Industry); Aventis Pharmaceuticals (Industry); GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 47; 104864-450
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2009-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Topotecan; Docetaxel

INTERVENTIONS:
Drug: Topotecan
Drug: Docetaxel

SUMMARY:
In this trial we will evaluate and compare the efficacy and toxicity of oral topotecan with intravenous docetaxel in the second-line treatment of patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be randomly assigned to one of two treatment arms:

* Topotecan
* Docetaxel

For ever 2 patients treated, 1 will receive treatment A (Topotecan) and 1 will receive treatment B (Docetaxel). The study is not blinded so both the patient and the doctor will know which treatment has been assigned.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Relapsed or Progressive Disease
* Stage IIIB (not candidate for combined modality) or IV
* No more than one prior chemotherapy regimen
* Able to perform activities of daily living without assistance
* Measurable disease outside of radiation port
* Adequate bone marrow, liver and kidney function
* Must understand study and sign informed consent prior to enrollment

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Prior treatment with Topotecan or Docetaxel
* Uncontrolled brain metastases
* Moderate peripheral neuropathy

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2000-11; Primary Completion 2005-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate

SECONDARY OUTCOMES:
Time to Progression
Overall survival
Overall toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Howard A. Burris, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States

REFERENCES:
- [Result] Jones S, Thompson D, Barton J, Patton J, Shipley D, Greco FA, Spigel D, Infante J, Burris HA 3rd. A randomized phase II trial of oral topotecan versus docetaxel in the second-line treatment of non-small-cell lung cancer. Clin Lung Cancer. 2008 May;9(3):154-9. doi: 10.3816/CLC.2008.n.023. PMID 18621625
- See also: Published article in Clinical Lung Cancer — http://cigjournals.metapress.com/content/478070h11q4u4l0g/fulltext.pdf